CLINICAL TRIAL: NCT03223519
Title: Double-blind, Randomized, Placebo-controlled, Single-center, Exploratory Clinical Trial to Investigate Safety and Efficacy of COMBOPROFEN for Treatment of Muscular Pain Associated With DOMS.
Brief Title: COMBOPROFEN for Treatment of Muscular Pain Associated With Delayed Onset Muscle Soreness (DOMS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spherium Biomed (Industry)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JAN12006-09; 2016-003139-39 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Delayed Onset Muscle Soreness, DOMS
Keywords: DOMS; Exercise; Ibuprofen; Magnesium; Vitamin C; Muscle pain
MeSH Terms: conditions — Motor Activity; Myalgia | interventions — Ibuprofen; Magnesium; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Comboprofen (Experimental): Triple combination of Ibuprofen, Magnesium and Vitamin C.
  Interventions: Drug: Comboprofen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- Magnesium (Active Comparator)
  Interventions: Drug: Magnesium
- Vitamin C (Active Comparator)
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Comboprofen — Triple combination of Ibuprofen, Magnesium and Vitamin C Powder for oral solution administered TID for 3 days
  Arms: Comboprofen
Drug: Placebo — Powder for oral solution administered TID for 3 days
  Arms: Placebo
Drug: Ibuprofen — Powder for oral solution administered TID for 3 days
  Arms: Ibuprofen
Drug: Magnesium — Powder for oral solution administered TID for 3 days
  Arms: Magnesium
Drug: Vitamin C — Powder for oral solution administered TID for 3 days
  Arms: Vitamin C

SUMMARY:
The study is designed as a proof of concept, single-center, randomized, double-blind, placebo controlled study to assess the safety and efficacy of Comboprofen (Ibuprofen + Magnesium + Vitamin C) compared to placebo, Ibuprofen, Magnesium and Vitamin C monotherapies in the treatment of Delayed Onset Muscle Soreness (DOMS).

DETAILED DESCRIPTION:
The study is designed as a proof of concept, single-center, randomized, double-blind, placebo controlled study to assess the safety and efficacy of Comboprofen (Ibuprofen + Magnesium + Vitamin C) compared to placebo, Ibuprofen, Magnesium and Vitamin C monotherapies in the treatment of Delayed Onset Muscle Soreness (DOMS).

Healthy volunteers will be recruited to undergo a controlled exercise test designed to induce DOMS in lower limbs. Subjets reporting sufficient pain intensity while walking in an 11-point Numerical Rating Scale (NRS) 24h or 48 h after exercise will be randomized to receive treatment with Comboprofen, placebo, ibuprofen, magnesium or vitamin c three times a day (TID) for 3 days.

Once a subject is randomized the duration of participation will be 7 days. Subjects will be housed in the clinic for the first 24 hours of dosing. Pain intensity while standing up and sitting down and while walking will be assessed throughout the study using an 11-point (0-10) Numeric Rating Scale (NRS). Maximal isometric force, muscle damage and inflammatory markers will be also assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, 18-45 years (inclusive) of age at the time of enrolment.
2. Body weight within normal range (Quetelet's index between 19 and 30) expressed as weight (kg) / height (m2).
3. Normal clinical records and physical examination.
4. No known musculoskeletal pathology.
5. Laboratory tests (hematology and biochemistry) within the range of normal values, according to the Biochemistry laboratory reference values of the 'Hospital de la Santa Creu i Sant Pau'. Variations may be admitted according to the clinical criteria of the CIM (Centre d'Investigació de Medicaments)-Sant Pau.
6. Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP (Systolic blood pressure) between 100-140 mm Hg/ DBP (Diastolic blood pressure) between 50-90 mm Hg / Heart rate between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
7. To be able to understand the nature of the study and comply with all their requirements.
8. Free acceptance to participate in the study by obtaining signed informed consent form approved by the CREC (Clinical Research Ethic Committee).
9. Not engaged in regular lower extremity fitness activities for more than 2 times per week for ≥ 2 consecutive weeks in the past 6 months before screening.

Exclusion Criteria:

1. History of alcohol dependence or drug abuse in the last 1 year or daily consumption of alcohol > 40 g/day for men or 24 g/day for women.
2. Heavy consumer of stimulating beverages (>5 coffees, teas, chocolate or cola drinks per day) and grapefruit juice.
3. Background of allergy, idiosyncrasy or hypersensitivity to drugs.
4. Intake of any medication within 4 days prior to induction of DOMS that could interfere with pain or muscle function, including over-the-counter products (including natural food supplements, vitamins and medicinal plants products), any source of Magnesium and Vitamin C and ionic and protein supplements.
5. Positive serology for hepatitis B, C or HIV.
6. Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological or neurological disease or other chronic diseases.
7. Twelve lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
8. Having undergone major surgery during the previous 6 months.
9. Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc.) from 6 months prior to drug administration.
10. Participation in another clinical trial during the 3 months preceding the drug administration.
11. Donation of blood during the 4 weeks preceding the drug administration.
12. Acute illness four weeks before drug administration.
13. Clinically significant abnormal laboratory values (as determined by the PI) at the screening evaluation.
14. Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract
15. Positive results of the drugs at screening period, at visit 2 before starting induction of DOMS or at visit 3 before starting treatment. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the PI).
16. Subjects who have been engaged in regular lower extremity fitness activities within 4 days prior to visit 2 (induction of DOMS).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference (SPID) while standing up and sitting down. | Over the first 72 hours after start of treatment.

SECONDARY OUTCOMES:
Summed Pain Intensity Difference (SPID) while standing up and sitting down and while walking. | Over the first 24, 48 and 72 hours after start of treatment.
Percentage of subjects achieving at least 50% or 70% reduction in pain intensity vs baseline while standing up and sitting down and while walking. | Over the first 24, 48 and 72 hours after start of treatment.
Percentage os subjects achieving at least 50% or 70% reduction in pain intensity vs baseline while climbing 9-step flight of stairs and while descending 9-step flight of stairs. | Over the first 24 and 72 hours after start of treatment.
Time to reduction of at least 50% or 70% pain intensity vs baseline while standing up and sitting down and while walking. | Over the first 72 hours after start of treatment.
Pain intensity difference (PID) while standing up and sitting down and while walking from baseline. | At 24 hours, 48 hours, 72 hours and 6-7 days after start of treatment.
Pain intensity difference (PID) while ascending and descending 9-step flight of stairs from baseline. | At 24 hours, 72 hours and 6-7 days after start of treatment.
Change in pain intensity while descending 9-step flight of stairs from baseline. | At 24 hours, 72 hours and 6-7 days after start of treatment.
Percentage of subjects achieving at least 80% or 100% recovery of baseline maximal isometric force. | At 24 hours, 72 hours and 6-7 days after start of treatment.
Change in perception of loss of strength induced by Comboprofen from baseline. | At 24 hours, 72 hours and 6-7 days after start of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain